CLINICAL TRIAL: NCT02664077
Title: A Phase III Randomized Placebo-Controlled Study Evaluating Regorafenib Following Completion of Standard Chemotherapy for Patients With Stage III Colon Cancer
Brief Title: A Study Evaluating Regorafenib Following Completion of Standard Chemotherapy for Patients With Colon Cancer
Acronym: ARGO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the significantly lower than expected accrual it was impossible to evaluate the endpoint in a timely fashion.
Sponsor: NSABP Foundation Inc (Network)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NSABP C-13; 17808 (Other: Bayer HealthCare Pharmaceuticals)
Record Dates: First submitted 2015-12-04; First posted 2016-01-26 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Stage III (IIIB or IIIC) Colon Cancer
Keywords: NSABP; Colon cancer; Regorafenib; Stage III; Adjuvant therapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Regorafenib (Experimental): Patients receive regorafenib orally once daily for 21 days of a 28 day cycle for a total of 26 cycles.
  Interventions: Drug: Regorafenib
- Group 2: Placebo (Placebo Comparator): Patients receive placebo orally once daily for 21 days of a 28 day cycle for a total of 26 cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Regorafenib — 3 tablets once a day by mouth for 21 consecutive days of 28 day cycle for 26 cycles
  Other Names: Stivarga
  Arms: Group 1: Regorafenib
Drug: Placebo — 3 tablets once a day by mouth for 21 consecutive days of 28 day cycle for 26 cycles
  Arms: Group 2: Placebo

SUMMARY:
This study is a randomized, double-blind, post-chemotherapy, adjuvant phase III clinical trial. The primary aim of this study is to determine the value of regorafenib in improving disease-free survival (DFS). Patients with Stage III (IIIB or IIIC) colon cancer as defined by the 7th Edition of the American Joint Committee on Cancer (AJCC) Cancer Staging Manual are randomized 1:1 to placebo or the experimental agent regorafenib following completion of at least four months of standard adjuvant therapy (e.g., 5-fluorouracil, leucovorin, oxaliplatin (FOLFOX) , capecitabine, oxaliplatin (CapeOx), and other).

DETAILED DESCRIPTION:
The primary aim of this study is to determine the value of regorafenib in improving DFS. The secondary aims are to evaluate the dose tolerance and long term toxicity of two years of regorafenib following standard adjuvant therapy, and to evaluate the effect of the use of regorafenib in overall survival (OS).

Eligible patients in this double-blind study will be randomized to take either regorafenib 120 mg or placebo orally, once daily for 21 consecutive days of a 28 day cycle for 26 cycles (2 years).

Accrual for this study will be approximately 1118 randomized patients. These 1118 patients will provide approximately 313 DFS events at the time of primary analysis. An initial futility analysis will be performed when 312 patients have been on study at least 3 months. The decision to continue the trial will be determined by success of both early stopping endpoints defined as follows:

* The toxicity profile of regorafenib compared to placebo is acceptable.
* The regorafenib regimen is tolerable for prolonged administration.

An estimated compliance rate of 60% at 6 months for regorafenib will be required for continuation of the study.

If toxicity is acceptable and compliance with regorafenib is at least 60% nominally, then accrual will continue.

The second futility analysis will be conducted when approximately 67 DFS events are observed. Trial conduct and accrual will continue unless the primary endpoint (DFS) trends too far in the opposite direction (hazard ratio greater than or equal to 1.1).

Toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

NSABP C-13 will include a Behavioral and Health Outcomes correlative science component. A C-13 Quality of Life (QOL) questionnaire will be administered at baseline (after consent and prior to randomization) and at 3 months, 6 months, 12 months, 18 months, 24 months, and 30 months.

Submission of blood samples for C-13 correlative science studies will be a study requirement for all patients. Submissions will also include archived primary tumor tissue from the resected colon primary. Blood samples for pharmacokinetics (PK) will be collected on Day 15 of Cycle 1 and Day 15 of Cycle 2, with additional blood samples for biomarkers collected at various time points for future analysis.

ELIGIBILITY:
Inclusion Criteria:

* The Eastern Cooperative Oncology Group (ECOG) performance status must be 0-1
* There must be histologic confirmation of high risk, adenocarcinoma of the colon defined as AJCC 7th Edition Stage IIIB or IIIC.
* The patient must have had an en bloc complete gross resection of tumor (curative resection) by open laparotomy or laparoscopically-assisted colectomy. The distal extent of the tumor must have been greater than or equal to 12 cm from the anal verge. (Patients who have had a two-stage surgical procedure to first provide a decompression colostomy and then in a later procedure to have a surgical resection are eligible.)
* Imaging (positron emission tomography/computed tomography (PET/CT) scan, CT scan, or magnetic resonance imaging (MRI)) of chest, abdomen, and pelvis must be performed within 90 days prior to randomization and must demonstrate no evidence of metastatic disease. If findings noted in imaging study reports are equivocal, the determination of whether or not the findings represent metastatic disease will be at the investigator's discretion.
* The patient must be able to swallow oral medication.
* The patient must have completed at least 4 months of adjuvant chemotherapy (i.e., FOLFOX, CapeOx, or other, such as 5-fluorouracil, leucovorin, oxaliplatin (FLOX), 5-fluorouracil/leucovorin (5FU/LV), capecitabine).
* The interval between completion of standard adjuvant chemotherapy and randomization must be less than or equal to 60 days.
* Blood counts performed within 28 days prior to randomization must meet the following criteria:

  * Absolute neutrophil count (ANC) must be greater than or equal to 1500/mm3;
  * platelet count must be greater than or equal to 100,000/mm3; and
  * hemoglobin must be greater than or equal to 9 g/dL.
* The following criteria for evidence of adequate hepatic function performed within 4 weeks prior to randomization must be met:

  * total bilirubin must be less than or equal to 1.5 x upper limit of normal (ULN); and
  * alkaline phosphatase must be less than or equal to 2 x ULN; and
  * Asparate aminotransferase (AST) and alanine aminotransferase (ALT) must be less than or equal to 2 x ULN for the lab. (Note: If AST and/or ALT greater than ULN, serologic testing for Hepatitis B and C must be performed and results must be negative.)
* Lipase performed within 28 days of randomization must be less than or equal to 1.5 x ULN for the lab.
* Serum creatinine performed within 28 days of randomization must be less than or equal to 1.5 x ULN for the lab.
* Urinalysis dipstick for urinary protein performed within 28 days prior to randomization must be 0-1+ protein. If urine dipstick result is greater than or equal to 2+ protein, a 24-hour urine protein must be less than 1.0 g/24 hours.
* Glomerular filtration rate (GFR) must be greater than or equal to 30 mL/min/1.73 m2 according to the Modified Diet in Renal Disease (MDRD) abbreviated formula.
* International normalized ratio of prothrombin time must be less than or equal to 1.5 times the ULN. Patients who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no underlying abnormality in coagulation parameters exists per medical history.
* Patients (male or female) of reproductive potential must agree to use an effective method of contraception (as discussed with treating physician) from the time consent is signed, during study therapy, and for at least 90 days after the last dose of study therapy.
* Patients with prior malignancies are eligible if they have been disease-free for at least 5 years and are deemed by their physician to be at low risk for recurrence. Patients with squamous or basal cell carcinoma of the skin, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum that have been effectively treated are eligible, even if these conditions were diagnosed within 5 years of randomization.

Exclusion Criteria:

* Isolated, distant, or non-contiguous intra-abdominal metastases, even if resected.
* Colon cancer other than adenocarcinoma (e.g., sarcoma, lymphoma, carcinoid).
* Prior history of invasive adenocarcinoma of colon or rectum.
* Patients with active autoimmune disease. (Patients with endocrine autoimmune diseases requiring replacement therapy alone are allowed.)
* Gastroduodenal ulcer(s) determined by endoscopy to be active.
* Any malabsorption condition.
* Known history of human immunodeficiency virus (HIV) infection or chronic or active hepatitis B or hepatitis C requiring treatment with antiviral therapy.
* Any concomitant systemic therapy or radiation therapy initiated for this malignancy.
* Active infection, or chronic infection requiring chronic suppressive antibiotics.
* Persistent CTCAE v4.0 greater than or equal to grade 2 diarrhea regardless of etiology.
* Know history of allografts (including corneal transplant).
* Chronic daily treatment with corticosteroids with a dose of greater than or equal to 10 mg/day methylprednisolone equivalent (excluding inhaled steroids), or any other immunosuppressive drugs.
* Any significant bleeding (greater than or equal to grade 3, hemorrhage) that is not related to the primary colon tumor within 6 months before randomization.
* Any of the following cardiac conditions:

  * documented New York Heart Association (NYHA) Class III or IV congestive heart failure;
  * myocardial infarction within 6 months prior to randomization;
  * unstable angina (angina symptoms at rest) within less than or equal to 3 months prior to randomization; and
  * clinically significant symptomatic arrhythmia despite anti-arrhythmic therapy.
* Uncontrolled blood pressure (systolic pressure greater than 150 mmHg or diastolic pressure greater than 90 mmHg on repeated measurements).
* Symptomatic brain or meningeal tumors.
* Patients with seizure disorder requiring medication.
* Presence of non-healing wound, non-healing ulcer, or bone fracture.
* Symptomatic interstitial lung disease or definitive evidence of interstitial lung disease described on CT scan, MRI, or chest x-ray in asymptomatic patients; dyspnea at rest requiring current continuous oxygen.
* Arterial or venous thrombotic or embolic events such as cerebral vascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before randomization (except for adequately treated catheter-related venous thrombosis occurring within 6 months before randomization).
* Symptomatic peripheral ischemia.
* Psychiatric or addictive disorders or other conditions or unresolved toxicities of prior therapy greater than grade 2 that, in the opinion of the investigator, would preclude the patient from meeting the study requirements, or interfere with interpretation of study results.
* Pregnancy or lactation at the time of study entry. (Note: Pregnancy testing must be performed within 14 days prior to randomization according to institutional standards for women of childbearing potential.)
* Major surgery (including ostomy reversal), open biopsy or significant trauma injury, within 28 days prior to randomization.
* Anticipation of need for major surgical procedures during the course of study.
* Known hypersensitivity to study drug, study drug classes or excipients of the formulation.
* Use of any vascular endothelial growth factor (VEGF) targeted therapy or previous use of regorafenib.
* Patients taking strong inducers or inhibitors of cytochrome P450 3A4 (CYP3A4) who cannot interrupt therapy from the time the C-13 consent is signed through 30 days after the last dose of study therapy.
* Patients taking herbal remedies (e.g., St. John's Wort [Hypericum perforatum]) who cannot interrupt therapy from the time the C-13 consent is signed through 30 days after the last dose of study therapy.
* Use of immune modulators and/or any immunosuppressive drugs.
* Use of any investigational agent within 28 days of randomization.
* Patients receiving erythropoiesis-stimulating agents or other hematopoietic growth factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Disease-free survival (DFS) - time from randomization until first colon cancer recurrence, second primary colon cancer, or death due to any cause. | Beginning at day 1 of cycle 3 (each cycle = 28 days) and every 6 months until study closure about 10 years
  To determine whether treatment with regorafenib following adjuvant therapy improves disease-free survival (DFS) in patients with Stage IIIB or IIIC colon cancer

SECONDARY OUTCOMES:
Overall Survival (OS) - time from randomization until death from any cause. | Day 1 of every cycle of chemotherapy then 30 days post study therapy, then every 6 months (years 3-5) then yearly (years 6 & 7)
  Determine the overall Survival
Toxicity - frequency and severity of adverse events categorized using the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) | Every study visit through 30 days following study therapy
  Evaluate toxicity associated with study therapy
Compliance - Time to discontinuation of study therapy. | Every study visit through discontinuation of study therapy, assessed for up to 24 months
  Evaluate the overall tolerability and compliance with study therapy
Correlative Science - Biomarker evaluations | Before randomization, prior to beginning Cycle 6, every 6 months through year 5, and at the end of study therapy (maximum of 2 years).
  Explore molecular and genetic correlatives for the degree of benefit from regorafenib
Correlative Science - Pharmacokinetics - Plasma regorafenib concentrations | Day 15 of Cycle 1 and Cycle 2 of study therapy.
  Evaluation of exposure to regorafenib
Correlative Science - Pharmacodynamics | Day 15 of Cycle 1 and Cycle 2 of study therapy.
  Evaluation of relationship between plasma concentrations and/or dose, efficacy, or adverse events
Compare the symptoms experienced by patients receiving regorafenib to patients receiving placebo during treatment as measured by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Baseline, 3 months, 6 months, 12 months, 18 months, 24 months and 6 months after discontinuation of protocol therapy
  Severity of treatment related symptoms experienced by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation
Locations (51):
- United States (51):
  - St. Joseph Hospital of Orange, Orange, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Colorado Cancer Research Program, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Care Specialists of Illinois - Decatur Memorial Hospital, Decatur, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Norton Cancer Institute, Norton Healthcare Pavilion, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Berkshire Medical Center Cancer and Infusion Center, Pittsfield, Massachusetts
  - Breslin Cancer Center, Lansing, Michigan
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Nevada Cancer Research Foundation, Inc., Las Vegas, Nevada
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Waverly Hematology Oncology, Cary, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Margaret R. Pardee Memorial Hospital, Hendersonville, North Carolina
  - First Health of the Carolinas Cancer Center, Pinehurst, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - James Cancer Hospital and Solove Research Institute at the Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Abington Hospital -Jefferson South, Abington, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Reading Hospital - McGlinn Cancer Institute, West Reading, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - McLeod Cancer Center for Treatment and Research, Florence, South Carolina
  - Wellmont Medical Associates Oncology and Hematology, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Green Bay Oncology, Ltd. - St. Vincent Hospital, Green Bay, Wisconsin